CLINICAL TRIAL: NCT00218855
Title: A Phase 3 Study With Randomization to Melphalan/Prednisone/Thalidomide Versus Melphalan/Prednisone/Placebo to Patients With Previously Untreated Multiple Myeloma
Brief Title: Thalidomide to Patients With Previously Untreated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other); Nordic Myeloma Study Group, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMSG #12; NFR 90000288
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Phase 3, randomised, double blind study; thalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: thalidomide; Drug: placebo
- B (Active Comparator)
  Interventions: Drug: thalidomide; Drug: placebo

INTERVENTIONS:
Drug: thalidomide — tablets thalidomide start 100 mg x 2 escalating to 200 mg x 2 until plateau phase. Maintenance 100 mg x 2 until relapse. The same procedure is repeated by first relapse.
  Other Names: thalidomide, Talix
Drug: placebo — 100 mg x 2 mg tablets escalating to 200 mg x 2 until plateau phase. Maintenance 100 mg x 2 until relapse. This procedure is repeated by first relapse.
  Other Names: no other names

SUMMARY:
The purpose of this study is to test the effect of thalidomide in patients with multiple myeloma. The patients receive either thalidomide or a placebo tablet (neither patient nor doctor know which of these are given) in addition to the ordinary chemotherapeutic drug against multiple myeloma. We will find out for how long time the patients will stay free of the disease and for how long time they will live, and can evaluate whether thalidomide is a beneficial drug against this disease.

DETAILED DESCRIPTION:
Thalidomide has recently emerged as an effective treatment for patients with myeloma refractory to conventional chemotherapy. So far only limited experience is available on thalidomide for newly diagnosed myeloma. Therefore the Nordic Myeloma Study Group decided to perform a trial comparing traditional melphalan-prednisone therapy with melphalan-prednisone + thalidomide/placebo. The study design is a multicentre double-blind randomised placebo-controlled trial. Mainly patients >65 years of age will be included since patients <65 years will be treated with high dose chemotherapy with autologous stem cell support. The primary end-point is overall survival. Secondary end-points are quality of life, response rate, time to response, response duration and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma in need of treatment

Exclusion Criteria:

* Previous treatment against multiple myeloma
* Need of high dose chemotherapy with autologous stem cell support
* Women in fertile age
* Psychiatric disease or mental reduction leading to lack of cooperation
* Lack of consent
* Life expectancy below 3 months
* Active cancer of other etiology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2002-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
overall survival | october 2007

SECONDARY OUTCOMES:
Quality of life | october 2007
Time to response | october 2007
Frequency of response | october 2007
Time to progression | october 2007
Time to 2. response | october 2007
Frequency of 2. response | october 2007
Time to 2. progression | october 2007
Toxicity | october 2007
Time to definitive treatment failure | october 2007

CONTACTS AND LOCATIONS:
Overall Officials: Anders Waage, MD, Study Chair — Department of Haematology, St. Olavs hospital/NTNU, N-7006 Trondheim
Locations (1):
- Department of Haematology, St. Olavs hospital/NTNU, Trondheim, Norway

REFERENCES:
- [Result] Waage A, Gimsing P, Fayers P, Abildgaard N, Ahlberg L, Bjorkstrand B, Carlson K, Dahl IM, Forsberg K, Gulbrandsen N, Haukas E, Hjertner O, Hjorth M, Karlsson T, Knudsen LM, Nielsen JL, Linder O, Mellqvist UH, Nesthus I, Rolke J, Strandberg M, Sorbo JH, Wisloff F, Juliusson G, Turesson I; Nordic Myeloma Study Group. Melphalan and prednisone plus thalidomide or placebo in elderly patients with multiple myeloma. Blood. 2010 Sep 2;116(9):1405-12. doi: 10.1182/blood-2009-08-237974. Epub 2010 May 6. PMID 20448107